CLINICAL TRIAL: NCT04245891
Title: Neonatal Evaluation of Norepinephrine Infusion in Spinal Anesthesia for Cesarean Section
Acronym: NECS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 17.11.01
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Caesarean Section;Stillbirth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: boli of ephedrine phenylephrine (45μg/mL-3mg/mL) if the variation of MAP < 20% of baseline (MAP before spinal anaesthesia).
- Protocol group: continuous infusion of norepinepineprhine at 20 μg/mL, started at 0.05 μg/kg/min. The dosage of norepinephrine was then adjusted to maintain a variation in MAP < 20% of baseline. In case of failure, the use of a control group boli injection was possible.

SUMMARY:
This retrospective study aims to evaluate the fate of children born by cesarean section under spinal anesthesia with or without norepinephrine as vasopressor support for anesthesia. The main objective is to compare the initial Apgar score. The records of patients who received norepinephrine are compared to those without norepinephrine. To limit the biases of this type of study, the investigators will apply a propensity score that will include as a variable: age, ASA score, comorbidity, urgency. The patients analysed correspond to the period 2016-2017.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* Spinal Anesthesia for Cesarean Section

Exclusion Criteria:

* sub epidural cesarean section
* contraindication to spinal anesthesia (allergy, severe heart disease, coagulopathy)

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: women over 18 years of age who need a caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
lactate level | Just after the birth of the newborn baby
  The primary endpoint is the Umbilical Cord Lactate levels

SECONDARY OUTCOMES:
APGAR Score | 1, 5 and 10 minutes after birth
  APGAR Score
Umbilical Cord arterial PH | Just after the birth
  Umbilical Cord arterial PH
Umbilical Cord venous PH | Just after the birth
  Umbilical Cord venous PH
maternal arterial tension during cesarean section | 0, 5,10,15, 20 25, 30,35,40 minutes after spinal anesthesia
  maternal arterial tension during cesarean section
incidences of mother nausea and vomiting | from beginning to cesarean section end
  incidences of mother nausea and vomiting
use of vasopressors | from beginning to cesarean section end
  use of vasopressors

IPD SHARING:
Plan to Share IPD: No